CLINICAL TRIAL: NCT07354269
Title: Phase IV Clinical Study Comparing the Immunogenicity and Safety of a Single-dose Poliomyelitis Vaccine (Vero Cells), Inactivated, Sabin Strains (sIPV) in Adolescents and Adults Aged 7-50 Years Versus the Primary Immunization With DTaP-IPV-Hib Pentavalent Vaccine in Infants Aged 3 Months
Brief Title: Phase IV Clinical Study of sIPV Administration in Adolescent and Adult Populations
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-sIPV-4004
Record Dates: First submitted 2025-04-22; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-04

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis | interventions — diphtheria-tetanus-five component acellular pertussis-inactivated poliomyelitis -Haemophilus influenzae type b conjugate vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sIPV group (Experimental): adolescents or adults aged 7-50 years
  Interventions: Biological: sIPV
- DTaP-IPV-Hib group (Active Comparator): infants aged 3 months old
  Interventions: Biological: DTaP-IPV-Hib

INTERVENTIONS:
Biological: sIPV — one dose of sIPV administered via intramuscular injection
  Arms: sIPV group
Biological: DTaP-IPV-Hib — three doses of DTaP-IPV-Hib administered via intramuscular injection following the schedule of 3,4,5 months old
  Arms: DTaP-IPV-Hib group

SUMMARY:
The goal of this clinical study is to compare the immunogenicity and safety of one dose of sIPV in adolescents or adults aged 7-50 years with that of three doses of DTaP-IPV-Hib Pentavalent Vaccine in Infants Aged 3 Months

DETAILED DESCRIPTION:
This study adopts a single-center, open-label, controlled design, planning to recruit 180 healthy participants, including 60 adolescents aged 7-17 years, 60 adults aged 18-50 years, and 60 infants aged 3 months. After being screened and enrolled, adolescents and adults aged 7-50 years will receive one dose of sIPV (inactivated poliovirus vaccine, Sabin strain) on Day 0, while infants aged 3 months will receive three doses of the pentavalent vaccine (DTaP-IPV-Hib) at 3, 4, and 5 months of age. Approximately 2.5-3.0 milliliters of venous blood will be collected from all participants before vaccination and on Day 30 after the last vaccination for antibody testing and immunogenicity evaluation. Researchers will observe participants for adverse events (AEs) within 30 minutes post-vaccination on-site and use diary cards to collect solicited and unsolicited AEs from Day 0 to Day 7 and AEs from Day 8 to Day 30 post-vaccination. Additionally, serious adverse events (SAEs) will be collected from the start of the first vaccination until Day 30 after the last vaccination. For fertile participants, pregnancy events for female participants themselves or the partners of male participants aged 18-50 years will be collected during the study period and after the first vaccination through a combination of active follow-up by researchers and self-reporting by participants.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adolescents and adults aged 7-50 years, and healthy infants aged 3 months;
2. Participants and/or their guardians are able to understand and voluntarily sign the informed consent form (for participants aged 7-17 years, both the participant and their guardian need to sign);
3. Provide valid proof of identity;
4. Willing and able to comply with all visit schedules, sample collections, vaccinations, and other study procedures, and remain contactable throughout the study period;
5. Fertile participants and their sexual partners voluntarily adopt effective contraceptive measures from the signing of the informed consent form until 3 months after vaccination with the study vaccine, and have no plans to donate sperm or eggs.

Exclusion Criteria:

1. Known history of polio/polio infection.
2. Exposure or suspected exposure to pertussis, diphtheria, and tetanus within the past 30 days, such as having a confirmed case of pertussis or diphtheria in the household (applies to infants aged 3 months).
3. History of uncontrolled chronic or severe illnesses, including but not limited to cardiovascular disease, hematological disorders, liver and kidney diseases, digestive system diseases, respiratory diseases, malignant tumors, and history of major organ transplantation.
4. Presence of autoimmune diseases, immunodeficiency disorders (including but not limited to systemic lupus erythematosus, ankylosing spondylitis, autoimmune thyroid diseases, asplenia, functional asplenia, and HIV infection).
5. Abnormal coagulation function (such as coagulation factor deficiency, platelet abnormalities).
6. Premature birth (delivery before the 37th week of gestation) or low birth weight (birth weight <2500g), or history of asphyxiation, or history of neurological damage (applies to infants aged 3 months).
7. Severe congenital malformations, genetic defects, and malnutrition.
8. Current or past history of severe neurological diseases (epilepsy, convulsions or seizures [excluding a history of febrile seizures]) or psychiatric disorders, or family history of psychiatric disorders.
9. Acute exacerbations of various acute or chronic diseases within the past 3 days, or known or suspected active infections.
10. History of vaccination with any vaccine containing DTP, IPV, Hib components, or pneumococcal polysaccharide conjugate vaccine (applies to infants aged 3 months).
11. Received immunosuppressive or other immunomodulatory treatment for ≥14 days within the past 6 months (≥20mg/day of prednisone for those ≥18 years old, ≥2mg/kg/day for those <18 years old, or equivalent doses), cytotoxic treatment, or plans to receive such treatment during the study.
12. Received immunoglobulin or other blood products within the past 6 months, or plans to receive such treatment during the study.
13. Received other investigational drugs or vaccines within the past 30 days, or plans to receive such drugs or vaccines during the study.
14. Received live attenuated vaccines, nucleic acid vaccines within the past 14 days, or subunit or inactivated vaccines within the past 7 days.
15. Known allergy to any component of the study vaccine (inactivated poliovirus, 199 medium, glycine, sodium chloride, potassium chloride, calcium chloride, magnesium phosphate, disodium phosphate, monosodium phosphate [for adolescents and adults]; inactivated poliovirus, diphtheria toxoid, tetanus toxoid, pertussis toxoid, pertussis filamentous hemagglutinin, Haemophilus influenzae type b capsular polysaccharide, tetanus protein conjugate [for infants aged 3 months]).
16. Breastfeeding, pregnant, or planning to become pregnant within 3 months after vaccination in this study (applies only to adolescents and adults).
17. Axillary temperature >37.0°C before vaccination on the day of the planned vaccination with the study vaccine.
18. Unqualified physical examination results on the day of the planned vaccination with the study vaccine.
19. Skin injuries, inflammation, ulcers, rashes, scars, or other conditions at the intended injection site that may interfere with vaccination or observation of local reactions.
20. Any other factors deemed unsuitable for participation in the clinical study by the investigator.

Ages: 3 Months to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2026-04-11 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
The SCR of nab against three serotypes of polioviruses at day 30 after one dose of sIPV in participants aged 7-17 years | day 30 after the single dose vaccination
  SCR indicates seroconversion rate；nab indicates neutralizing antibody
The SCR of nab against three serotypes of polioviruses at day 30 after one dose of sIPV in participants aged 18-50 years | day 30 after the single dose vaccination
  SCR indicates seroconversion rate; nab indicates neutralizing antibody
The SCR of nab against three serotypes of polioviruses at day 30 after three doses of DTaP-IPV-Hib in infants aged 3 months | day 30 after the single dose vaccination
  SCR indicates seroconversion rates; nab indicates neutralizing antibody

SECONDARY OUTCOMES:
The frequency of adverse reactions within 30 days after vaccination in participants aged 7-50 years | 0-30 days after vaccination
The frequency of SAEs within 30 days after vaccination in participants aged 7-50 years | 0-30 days after vaccination
  SAE indicates serious adverse events
The frequency of adverse reactions within 30 days after vaccination in infants | 0-30 days after vaccination
The frequency of SAEs within 30 days after vaccination in infants | 0-30 days after vaccination
  SAE indicates serious adverse events
The SPR of antibody against PT at day 30 after three doses of DTaP-IPV-Hib in infants aged 3 months | day 30 after three doses of vaccination
  SPR indicates seropositivity rate; PT indicates pertussis toxin
The SCR of antibody against PT at day 30 after three doses of DTaP-IPV-Hib in infants aged 3 months | day 30 after three doses of vaccination
  SCR indicates seroconversion rates; PT indicates pertussis toxin
The SPR of antibddy against DT at day 30 after three doses of DTaP-IPV-Hib in infants aged 3 months | day 30 after three doses of vaccination
  SPR indicates seropositivity rate; DT indicates diphtheria toxin
The SCR of antibody against DT at day 30 after three doses of DTaP-IPV-Hib in infants aged 3 months | day 30 after three doses of vaccination
  SCR indicates seroconversion rate； DT indicates diphtheria toxin
The SPR of antibody against TT at day 30 after three doses of DTaP-IPV-Hib in infants aged 3 months | day 30 after three doses of vaccination
  SPR indicates seropositivity rate; TT indicates tetanus toxin
The SCR of antibody against TT at day 30 after three doses of DTaP-IPV-Hib in infants aged 3 months | day 30 after three doses of vaccination
  SCR indicates seroconversion rates; TT indicates tetanus toxin

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Longxi County Center for Disease Prevention and Control, Dingxi City, Dingxi, Gansu
  - Chengguan District Center for Disease Prevention and Control, Lanzhou City, Lanzhou, Gansu
  - Zhangye Center for Disease Prevention and Control, Zhangye, Gansu

IPD SHARING:
Plan to Share IPD: Undecided